CLINICAL TRIAL: NCT04225052
Title: A Randomized, Open-label, Single Dose, Crossover Clinical Trial to Compare the Safety and Pharmacokinetics of YHP1903 in Healthy Volunteers
Brief Title: Clinical Trial to Evaluate the Safety and Pharmacokinetics of YHP1903 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Collaborators: Chonbuk National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: YHP1903-101
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Healthy Volunteer
Keywords: Pharmacokinetics
MeSH Terms: interventions — Varenicline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group1 (Other): 16 subjects, Cross-over, Single dose of comparator on day1, Single dose of YHP1903 on day8
  Interventions: Drug: YHP1903; Drug: Champix
- Group2 (Other): 16 subjects, Cross-over, Single dose of YHP1903 on day1, Single dose of comparator on day8
  Interventions: Drug: YHP1903; Drug: Champix

INTERVENTIONS:
Drug: YHP1903 — YHP1903 Tab. 1mg
Drug: Champix — Comparator Champix Tab. 1mg

SUMMARY:
A randomized, open-label, single dose, crossover clinical trial to evaluate the safety and pharmacokinetics of YHP1903 in healthy volunteers

DETAILED DESCRIPTION:
32 healthy subjects wil be randomized one of 2 groups in the same ratio. Subjects in group 1 will be administered "comparator" and "YHP1903" by cross-over design on day1, 8.

Subjects in group 2 will be administered "YHP1903" and "comparator" by cross-over design on day1, 8.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male/female aged 19 to 55 with body mass index(BMI) between 18.5 and 30kg/m2
2. Acceptable medical history, physical examination, laboratory tests and EKG, during screening
3. Subjects who has signed a written informed consent voluntarily,prior to any procedure, using a form that is approved by the local Institutional Review Board after detail explanation of the purpose, contents, and characteristic of the drug

Exclusion Criteria:

1. History of clinically significant disease
2. Sitting blood pressure meeting the following criteria at screening:

   * 140 ≤ systolic blood pressure ≤90 (mmHg)
   * 90 ≤ diastolic blood pressure ≤ 60 (mmHg)
3. Have AST(SGOT) or/and ALT(SGPT) > 1.5 times of normal upper limit or Total bilirubin > 2.0 mg/dl at the time of screening
4. Volunteers considered not eligible for the clinical trial by the investigator
5. Administration of other investigational products within 6 month prior to the first dosing.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2020-01-08 (Actual); Study Completion 2020-01-14 (Actual)

PRIMARY OUTCOMES:
AUCt | 0-96 hours
  AUCt of Varenicline
Cmax | 0-96 hours
  Cmax of Varenicline

SECONDARY OUTCOMES:
AUCinf | 0-96 hours
  AUCinf of Varenicline
Tmax | 0-96 hours
  Tmax of Varenicline
t1/2 | 0-96 hours
  t1/2 of Varenicline

CONTACTS AND LOCATIONS:
Overall Officials: Mingul Kim, PhD, Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Chonbuk national university hospital, Jeonju, Jeollabuk-do, South Korea